CLINICAL TRIAL: NCT06483685
Title: Global Insights Into Therapeutic Radiopharmaceuticals Safety: A Comprehensive Analysis From the WHO Pharmacovigilance Database (RADIANTS)
Brief Title: Radiopharmaceuticals Analysis for Detailed Insights And INternational Tracking of Safety
Acronym: RADIANTS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 20240531; RADIANTS (Other: University Hospital Caen)
Record Dates: First submitted 2024-06-03; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Side Effect of Drug
Keywords: Pharmacovigilance; Adverse Drug Reactions; Nuclear Medicine; Radiotherapeutics
MeSH Terms: conditions — Neoplasms; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adverse Events with Radiopharmaceuticals drugs: Cases reported in the World Health Organization (WHO) of patients treated by Radiopharmaceuticals drugs with reported toxicity
  Interventions: Drug: Radiopharmaceuticals drugs

INTERVENTIONS:
Drug: Radiopharmaceuticals drugs — radiopharmaceuticals drugs included in the Anatomical Therapeutic Chemical (ATC) classification system.

SUMMARY:
Little is known about cancer therapy-related radiopharmaceuticals drugs safety. Here the investigators use VigiBase (http://www.vigiaccess.org/), the World Health Organization (WHO) database of individual safety case reports, to identify and describe cases of cancer therapy-related radiopharmaceuticals drugs.

DETAILED DESCRIPTION:
Radiopharmaceuticals drugs especially for therapeutic purposes are responsible of a wide range of side effects. The investigators use VigiBase, the World Health Organization (WHO) database of individual safety case reports, to identify cases of adverse drug reactions following treatment with radiopharmaceuticals drugs.

ELIGIBILITY:
Inclusion Criteria:

* cases reported in the World Health Organization (WHO) database of individual safety case reports (vigibase)

Exclusion Criteria:

* not related to radiopharmaceuticals

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases reported in the World Health Organization (WHO) database of individual safety case reports (vigibase) related to radiopharmaceuticals
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Toxicity of Radiopharmaceuticals drugs | Case reported in the World Health Organization (WHO) of individual safety case reports through study completion, an average 5 years
  Identification and report of toxicities of radiopharmaceuticals drugs. The research includes the report with MedDRA terms: System organ class (SOC), Preferred terms (PT), High level group term (HLGT), High level term (HLT)

SECONDARY OUTCOMES:
Individual safety case reports parameters | Through study completion, an average 5 years
  weight in kilograms, height in meters, age in years, country, date of report in years, co-medication in active ingredients name, sex (male / female), severity (yes or no), death reported (yes or no), reporter qualification, action taken with drug, outcome (recovered, not recovered, role of co-medication (suspect, concomittant, unknown), drugs doses (MegaBecquerels, milligrams, grams, international units, milliliters), route of administration. Date of suspected drug administration, Start date and end date of reported adverse events. Dechallenge of suspected drugs (yes , no, unknown), Rechallenge of suspected drugs (yes , no, unknown).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Vigne, PharmD, PhD, Principal Investigator — CHU de Caen Normandie
Locations (1):
- Caen Normandy University Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolladille C, Ederhy S, Ezine E, Choquet S, Nguyen LS, Alexandre J, Moslehi JJ, Dechartres A, Salem JE. Chimeric antigen receptor T-cells safety: A pharmacovigilance and meta-analysis study. Am J Hematol. 2021 Sep 1;96(9):1101-1111. doi: 10.1002/ajh.26259. Epub 2021 Jun 23. PMID 34057232
- [Background] Ladriere T, Faudemer J, Levigoureux E, Peyronnet D, Desmonts C, Vigne J. Safety and Therapeutic Optimization of Lutetium-177 Based Radiopharmaceuticals. Pharmaceutics. 2023 Apr 13;15(4):1240. doi: 10.3390/pharmaceutics15041240. PMID 37111725
- [Result] Vigne J, Chretien B, Bignon AL, Bouhier-Leporrier K, Dolladille C. [177Lu]Lu-DOTATATE peptide receptor radionuclide therapy-associated myeloid neoplasms: insights from the WHO pharmacovigilance database. Eur J Nucl Med Mol Imaging. 2022 Aug;49(10):3332-3333. doi: 10.1007/s00259-022-05833-6. Epub 2022 May 6. No abstract available. PMID 35513605